CLINICAL TRIAL: NCT06958016
Title: Investigation of the Role and Prognostic Value of Tryptase in Patients With Stable Coronary Artery Disease
Brief Title: Role of Tryptase Levels in Patients With Stable Coronary Artery Disease.
Acronym: TRY-CAD
Status: Recruiting | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Fotios Skoufis, Principal Investigator, University of Thessaly
Other Study IDs: 447
Record Dates: First submitted 2025-04-23; First posted 2025-05-06 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Chronic Coronary Syndrome
Keywords: chronic coronary syndrome; tryptase; biomarker; mast cell activation; plaque instability; prognosis; MACE; Stable Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Coronary Artery Disease Group: Patients with angiographically proven coronary artery stenosis >70%
- Non-coronary Artery Disease Group: Patients with angiographically proven coronary artery stenosis <70%

SUMMARY:
The aim of this study is to measure the levels of serum tryptase and correlate them with the severity of coronary artery disease in study population. In addition, it will evaluate the usability of tryptase levels as a prognostic biomarker for future cardiovascular events.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is the leading cause of death worldwide based on WHO' s latest review in 2019 with CAD being responsible for the 16% of them. The main feature of coronary artery disease is the accumulation of atherosclerotic plaque in the epicardial arteries whether obstructive or non-obstructive. CAD is further subclassified into Chronic Coronary Syndrome (CCS) and Acute Coronary Syndrome (ACS). Patients with CCS experience long and stable periods of myocardial ischemia. However, in the case of a plaque rapture these patients can turn into ACS patients. The objective of this study is to predict that sudden shifting of patients from CCS to ACS by associating the role of inflammation and its factors with cardiovascular events. In particular, it focuses on mast cell (MC) tryptase which provokes plaque instability in patients with CCS. Mast cells needs to be activated to release tryptase and their activation mechanism seems to be the bridging point between tryptase and coronary artery disease. Previous studies have shown that IgE levels, which is the most potent activator of MC, are found high in hyperlipidemic patients. In addition, oxidized LDL (Ox-LDL) is another MC activator.

In reference to the fact that there might be a correlation between tryptase and coronary plaque instability in patients with chronic coronary syndrome, the investigator propose an interventional study for the role of tryptase as a prognostic biomarker in patients with CCS by studying a large population of Greek subjects with CCS.

The study will be conducted on 2 patient population:

1. Patients without coronary artery disease (estimated stenosis <70%) - Control group
2. Patients with coronary artery disease (estimated stenosis >70%) - CAD group

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 - 85 years old.
* Clinical symptoms of angina which are classified based on the Canadian Cardiovascular Score (CCS score)
* Positive SPECT scan for myocardial ischemia

Exclusion Criteria:

* Acute Coronary Syndrome 4 weeks before the coronary catheterization
* Percutaneous Coronary Angioplasty
* Coronary Artery Bypass Graft
* Active symptoms of allergy (asthma, urticaria)
* Mastocytosis
* Hypereosinophilia
* Autoimmune disease
* Cancer
* Kidney failure
* Myelodysplastic Syndrome
* Denial of signing informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a multicentre study which take place at the military hospital 417 NIMTS, Athens and the Larissa University Hospital, Larissa. Participants from both locations are patients who are going to undergo percutaneous coronary intervention. These patients will enter the study after fulfiling the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2026-01-11 (Estimated); Study Completion 2027-01-11 (Estimated)

PRIMARY OUTCOMES:
Serum tryptase levels as a biomarker in CCS | Baseline
  Correlation of tryptase levels with Coronary Artery Disease gravity

SECONDARY OUTCOMES:
Tryptase and major cardiovascular evens | 12 months after the completion of recruitment
  Correlation of tryptase levels with possible major cardiovascular events (death, myocardial infarction)

CONTACTS AND LOCATIONS:
Overall Officials: Grigorios Giamouzis, PhD Medicine, Study Director — University of Thessaly
Locations (2):
- Greece (2):
  - 417 Military Hospital NIMTS, Athens, Attica
  - Larisa University Hospital, Larissa, Thessaly